CLINICAL TRIAL: NCT00002330
Title: A Randomized Study Comparing the Safety and Efficacy of Three Doses of Oral Ganciclovir to Intravenous Ganciclovir for the Maintenance Treatment of Cytomegalovirus Retinitis in People With AIDS
Brief Title: A Study of Two Forms of Ganciclovir in the Treatment of Cytomegalovirus (CMV) of the Eyes in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roche Global Development (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 059F; GANs2226
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To compare the time to progression of Cytomegalovirus (CMV) retinitis among each of three doses of oral ganciclovir, as well as to intravenous therapy, when given as maintenance for 26 weeks. To compare the safety and tolerance among oral doses of ganciclovir at the study doses, as well as to intravenous therapy, when administered as maintenance for 26 weeks.

DETAILED DESCRIPTION:
Patients who have received anti-CMV therapy with intravenous ganciclovir for at least 4 weeks that resulted in stable retinitis are randomized to receive one of three doses of oral ganciclovir or intravenous ganciclovir for 26 weeks of maintenance.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Topical and ophthalmic nucleoside analogues.

Patients must have:

* HIV positive.
* No more than two episodes of CMV retinitis progression (relapse resulting in reinduction with intravenous anti-CMV therapy) since the original retinitis diagnosis.
* Currently stable retinitis.

Prior Medication:

Allowed:

* Foscarnet prior to the 4 weeks of intravenous induction therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Persistent or clinically significant diarrhea, nausea, or abdominal pain.
* Severe odynophagia.
* Other gastrointestinal (GI) symptoms or uncontrolled GI disease.
* Active CMV disease of the GI tract (e.g., CMV colitis, CMV esophagitis).
* Ocular media opacities (corneal, lenticular, or vitreal) that prevent ophthalmologic retinal assessments.
* Dementia, decreased mentation, or other encephalopathic signs and symptoms that would preclude informed consent or study compliance.

Concurrent Medication:

Excluded:

* Acyclovir sodium (Zovirax) by any route other than topical.
* Valacyclovir.
* Brovavir.
* Vidarabine.
* Amantadine hydrochloride.
* Cytarabine.
* Idoxuridine.
* Ribavirin.
* Interferon.
* Foscarnet (non-nucleoside pyrophosphate analogue).
* CMV hyperimmune globulin.
* Soluble CD4.
* Trichosanthin (Compound Q).
* Imipenem-cilastatin.
* Isoprinosine.
* Levamisole.
* Other investigational drugs.

Patients with the following prior condition are excluded:

History of hypersensitivity to acyclovir or ganciclovir.

Prior Medication:

Excluded:

* More than three induction regimens with intravenous anti-CMV therapy.
* Any prior oral ganciclovir.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280

CONTACTS AND LOCATIONS:
Locations (36):
- United States (35):
  - Univ of Alabama at Birmingham / AIDS Outpatient Clinic, Birmingham, Alabama
  - McDowell Clinic, Phoenix, Arizona
  - Dr Ken Fisher, Phoenix, Arizona
  - Univ of Arizona / Health Science Ctr, Tucson, Arizona
  - East Bay AIDS Ctr, Berkeley, California
  - AIDS Clinical Research Ctr / UCLA Med Ctr, Los Angeles, California
  - UCSD Med Ctr / Pediatrics, San Diego, California
  - Davies Med Ctr, San Francisco, California
  - Mount Zion Med Ctr / UCSF, San Francisco, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Community Research Initiative, Coral Gables, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Margo Heath - Chiozzi, Honolulu, Hawaii
  - Univ of Maryland School of Medicine, Baltimore, Maryland
  - AIDS Clinical Trials Unit, St Louis, Missouri
  - HIV Wellness Ctr / Univ Med Ctr, Las Vegas, Nevada
  - Univ of New Mexico, Albuquerque, New Mexico
  - AIDS Wellness Clinic, Sante Fe, New Mexico
  - Dr Dorothy Friedberg, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - New York Hosp - Cornell Med Ctr, New York, New York
  - Univ of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Nalle Clinic, Charlotte, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp, Columbus, Ohio
  - Associates Med and Mental Health, Tulsa, Oklahoma
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Austin Infectious Disease Consultants, Austin, Texas
  - N Texas Ctr for AIDS & Clin Rsch, Dallas, Texas
  - Texas Tech Health Sciences Ctr, El Paso, Texas
  - Dr Daniel Barbero, Fort Worth, Texas
  - Infectious Diseases Association of Houston, Houston, Texas
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas
- Saint Paul's Hosp, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Lalezari J, Friedberg D, Bisset J, Giordano M, Hardy D, Robinson C. A comparison of the safety and efficacy of 3g, 4.5g and 6g doses of oral ganciclovir versus IV ganciclovir for maintenance treatment of CMV retinitis. Int Conf AIDS. 1996 Jul 7-12;11(2):226 (abstract no ThB305)